CLINICAL TRIAL: NCT03394430
Title: Comparison of Intranasal Midazolam or Dexmedetomidine on Epileptiform EEG During Sevoflurane Mask Induction in Children
Brief Title: Comparison of Midazolam or Dexmedetomidine on Epileptiform EEG During Sevoflurane Mask Induction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Yu Sun, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MDZ/DEX
Record Dates: First submitted 2017-12-17; First posted 2018-01-09 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-02

CONDITIONS: Inhalation Anesthesia
Keywords: sevoflurane; epileptiform EEG; midazolam; dexmedetomidine
MeSH Terms: interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Placebo Comparator)
  Interventions: Drug: Placebos
- Group B (Experimental)
  Interventions: Drug: Midazolam
- Group C (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Placebos — Patients in Group A receive intranasal normal saline before anesthesia. Anaesthesia was induced with 8% sevoﬂurane initially. Sevoflurane concentration decreased to 2% after intubation. An electroencephalogram was recorded before and during induction up to 10 min after the start of induction.
  Arms: Group A
Drug: Midazolam — Patients in Group B receive intranasal 0.25mg/kg midazolam before anesthesia. Anaesthesia was induced with 8% sevoﬂurane initially. Sevoflurane concentration decreased to 2% after intubation. An electroencephalogram was recorded before and during induction up to 10 min after the start of induction.
  Arms: Group B
Drug: Dexmedetomidine — Patients in Group C receive intranasal 1μg/kg dexmedetomidine before anesthesia. Anaesthesia was induced with 8% sevoﬂurane initially. Sevoflurane concentration decreased to 2% after intubation. An electroencephalogram was recorded before and during induction up to 10 min after the start of induction.
  Arms: Group C

SUMMARY:
Induction with high sevoﬂurane concentrations may trigger epileptiform electroencephalographic activity without motor or cardiovascular manifestations in healthy patients. No other symptoms were associated in this series, and only electroencephalographic monitoring allowed the diagnosis. Midazolam and dexmedetomidine are sedatives commonly used in children before surgery. Although the mechanisms are different, both have been reported in antiepileptic effects.

This study was designed to compare the effects between intranasal midazolam or dexmedetomidine on epileptiform EEG during sevoflurane mask induction in children. Anaesthesia was induced with 8% sevoﬂurane. The patients were randomly assigned to Group A (n=15, preoperative intranasal normal saline), Group B (n=15, preoperative intranasal 0.25mg/kg midazolam), and Group C (n=15, preoperative intranasal 1μg/kg dexmedetomidine). An electroencephalogram was recorded before and during induction up to 10 min after the start of induction.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-2
* Scheduled for general anesthesia

Exclusion Criteria:

* Patients with a history of neurological, mental illnes
* Patients with a history of congenital heart disease
* Patients with a history of allergies to related drugs

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
incidence of epileptiform EEG | 0 min after induction, up to 10 min
  EEG were visually analyzed off-line by a neurophysiologist familiar with anesthesia EEG and blinded to the randomization. EEG abnormalities related to epileptic features were classiﬁed according to the description of Vakkuri and Jaaskelainen, and the recommendations of Constant: spikes and spikes with slow wave complexes (SW), rhythmic polyspikes corresponding to waveforms appearing at regular intervals (RPS) and periodic epileptiform discharge (PED), which refers to periodic hypersynchronized complexes occurring bilaterally. These entire electroencephalographic phenomena were considered as epileptiform EEG if their duration was longer than three seconds.

SECONDARY OUTCOMES:
electroencephalographic changes | 0 min after induction, up to 10 min
  the delay between the start of induction and the ﬁrst changes in electroencephalographic activity (appearance of β, θ, or δ rhythms)
electroencephalographic changes | 0 min after induction, up to 10 min
  the occurrence of burst suppressions
electroencephalographic changes | 0 min after induction, up to 10 min
  duration of suppression period, i.e. the sum of the EEG silences.
hemodynamic changes | 1 min before induction
  blood pressure
hemodynamic changes | 1 min before induction
  heart rate
hemodynamic changes | during induction procedure
  blood pressure
hemodynamic changes | during induction procedure
  heart rate
hemodynamic changes | 2 min after induciton
  blood pressure
hemodynamic changes | 2 min after induciton
  heart rate
hemodynamic changes | 4 min after induciton
  blood pressure
hemodynamic changes | 4 min after induciton
  heart rate
hemodynamic changes | 6 min after induciton
  blood pressure
hemodynamic changes | 6 min after induciton
  heart rate
hemodynamic changes | 8 min after induciton
  blood pressure
hemodynamic changes | 8 min after induciton
  heart rate
hemodynamic changes | 10 min after induciton
  blood pressure
hemodynamic changes | 10 min after induciton
  heart rate
intubation time | 0 min after intubation
  from taking of the intubation device to successful intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital,Affililated to Shanghai Jiaotong University School of Medicine, Shanghai, China